CLINICAL TRIAL: NCT06912035
Title: EFFICACY OF DIACEREIN ADDITION ON INTERLEUKIN-1Β, HS-CRP, TNF-Α LEVELS AND GLYCEMIC CONTROL IN UNCONTROLLED TYPE 2 DIABETES MELLITUS PATIENTS AT DR. MOHAMMAD HOESIN GENERAL HOSPITAL PALEMBANG
Brief Title: Efficacy of Diacerein Supplementation on Interleukin-1β, Hs-CRP, TNF-α Levels and Glycemic Control in Uncontrolled Type 2 Diabetes Mellitus Patients at Dr. Mohammad Hoesin General Hospital Palembang
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitas Sriwijaya (Other)
Collaborators: Indonesia Endowment Fund for Education (LPDP), Ministry of Finance Republik of Indonesia (Unknown)
Responsible Party: Principal Investigator, Yulianto Kusnadi, Dr. dr. Yulianto, SpPD, K-EMD, Universitas Sriwijaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DP0403/DXVIII0608/ETIK007/2025
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Uncontrolled Diabetes; Diabetes Mellitus Type 2
Keywords: Diacerein; Diabetes Mellitus Type 2; Uncontrolled Diabetes; Interleukin-1β; hs-CRP; TNF-α
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — diacerein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diacerein 50 mg capsules (Experimental): The patients were given a capsule containing Diacerein 50 mg twice a day
  Interventions: Drug: Diacerein 50 mg Capsule
- Placebo (Placebo Comparator): Patients received placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diacerein 50 mg Capsule — The patients received diacerein capsules
  Arms: Diacerein 50 mg capsules
Drug: Placebo — Patients received placebo capsules
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if diacerein supplementation can help improve inflammation and glycemic control in adults with uncontrolled type 2 diabetes. It will also study the safety and tolerability of diacerein. The main questions it aims to answer are:

* Does diacerein lower levels of inflammatory markers like interleukin-1β, hs-CRP, and TNF-α?
* Does diacerein improve blood sugar control?
* What side effects or problems do participants have when taking diacerein?

Researchers will compare diacerein to a placebo (a look-alike substance with no active drug) to see if it works better for managing type 2 diabetes.

Participants will:

* Be adults aged 40-60 with uncontrolled type 2 diabetes
* Take either diacerein or a placebo every day for 12 weeks
* Visit the clinic for blood tests and monitoring at the beginning and end of the trial
* Be evaluated for side effects and medication adherence]

DETAILED DESCRIPTION:
The study aimed to evaluate the efficacy of diacerein supplementation compared to placebo towards interleukin-1β, hs-CRP, TNF-α levels and glycemic control in uncontrolled type 2 diabetes mellitus patients. The current study was designed as a single-center double-blind randomized controlled clinical trial. The participants were voluntarily recruited 40-60 years old with uncontrolled type 2 diabetes mellitus. Participants were randomized into two groups receiving diacerein add-on therapy or placebo. Evaluations were conducted for side effects and adherence. towards Interleukin-1β, hs-CRP, TNF-α levels and glycemic control were evaluated at the beginning and at the end of the 12 weeks trial for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with uncontrolled type 2 diabetes mellitus who are receiving treatment at Dr. Mohammad Hoesin General Hospital, Palembang.
2. Male and female patients aged 40-59 years.
3. Willing to participate in the study by signing the informed consent form.

Exclusion Criteria

1. Pregnant or breastfeeding.
2. History of allergy to medications containing rhein.
3. Severe liver disorders.
4. Chronic kidney disease.
5. Malignancy.
6. Currently receiving hormone replacement therapy.
7. Autoimmune diseases.
8. Severe bacterial infection.
9. Osteoarthritis.
10. Use of other anti-inflammatory drugs within the past 2 weeks.

Drop-out Criteria

1. Patients who discontinue medication for more than 2 weeks.
2. Death.
3. Occurrence of serious adverse drug reactions requiring discontinuation of the medication.
4. Loss to follow-up.

Ages: 60 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | [Time frame: From enrollment to the end of the treatment at 12 weeks]
  To determine the effectiveness of adding diacerein compared to placebo towards Interleukin-1β, hs-CRP, TNF-α levels and glycemic control in uncontrolled type 2 diabetes mellitus patients.

SECONDARY OUTCOMES:
Secondary Outcome | [Time frame: From enrollment to the end of the treatment at 12 weeks]
  To analyze the difference in levels of HbA1C and fasting plasma glucose (FPG) before and after the addition of diacerein in patients with uncontrolled diabetes mellitus.
Secondary Outcome | [Time frame: From enrollment to the end of the treatment at 12 weeks]
  To analyze the difference in levels of Interleukin-1β before and after the addition of diacerein in patients with uncontrolled diabetes mellitus.
Secondary Outcome | [Time frame: From enrollment to the end of the treatment at 12 weeks]
  To analyze the difference in levels of hs-CRP before and after the addition of diacerein in patients with uncontrolled diabetes mellitus.
Secondary Outcome | [Time frame: From enrollment to the end of the treatment at 12 weeks]
  To analyze the factors associated with changes in serum interleukin-1β, hs-CRP, TNF-α and glycemic control before and after the addition of diacerein in patients with uncontrolled type 2 diabetes mellitus.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Sriwijaya, Palembang, South Sumatera, Indonesia

REFERENCES:
- [Background] Tres GS, Fuchs SC, Piovesan F, Koehler-Santos P, Pereira FDS, Camey S, Lisboa HK, Moreira LB. Effect of Diacerein on Metabolic Control and Inflammatory Markers in Patients with Type 2 Diabetes Using Antidiabetic Agents: A Randomized Controlled Trial. J Diabetes Res. 2018 Apr 2;2018:4246521. doi: 10.1155/2018/4246521. eCollection 2018. PMID 29805981
- [Background] Cardoso CRL, Leite NC, Carlos FO, Loureiro AA, Viegas BB, Salles GF. Efficacy and Safety of Diacerein in Patients With Inadequately Controlled Type 2 Diabetes: A Randomized Controlled Trial. Diabetes Care. 2017 Oct;40(10):1356-1363. doi: 10.2337/dc17-0374. Epub 2017 Aug 17. PMID 28818994
- [Background] Villar MM, Martinez-Abundis E, Preciado-Marquez RO, Gonzalez-Ortiz M. Effect of diacerein as an add-on to metformin in patients with type 2 diabetes mellitus and inadequate glycemic control. Arch Endocrinol Metab. 2017 Mar-Apr;61(2):188-192. doi: 10.1590/2359-3997000000242. Epub 2017 Feb 13. PMID 28225996
- [Background] Jangsiripornpakorn J, Srisuk S, Chailurkit L, Nimitphong H, Saetung S, Ongphiphadhanakul B. The glucose-lowering effect of low-dose diacerein and its responsiveness metabolic markers in uncontrolled diabetes. BMC Res Notes. 2022 Mar 4;15(1):91. doi: 10.1186/s13104-022-05974-9. PMID 35246243